CLINICAL TRIAL: NCT01828112
Title: A Phase III, Multicenter, Randomized, Open-label Study of Oral LDK378 Versus Standard Chemotherapy in Adult Patients With ALK-rearranged (ALK-positive) Advanced Non-small Cell Lung Cancer Who Have Been Treated Previously With Chemotherapy (Platinum Doublet) and Crizotinib
Brief Title: LDK378 Versus Chemotherapy in ALK Rearranged (ALK Positive) Patients Previously Treated With Chemotherapy (Platinum Doublet) and Crizotinib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2303; 2012-005637-36 (EudraCT Number)
Record Dates: First submitted 2013-04-02; First posted 2013-04-10 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; ALK; LDK378; Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; lung cancer; lung adenocarcinoma; Non small cell lung carcinoma; Non small cell lung cancer; NSCLC; chemotherapy; ALK-positive; ALK-rearranged advanced non-small cell lung cancer; crizotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — ceritinib; Pemetrexed; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ceritinib (Experimental): Ceritinib 750 mg
  Interventions: Drug: Ceritinib
- Chemotherapy (Active Comparator): Chemotherapy as determined by BIRC
  Interventions: Drug: Pemetrexed; Drug: Docetaxel

INTERVENTIONS:
Drug: Ceritinib — Ceritinib was the investigational treatment and was provided as 150 mg hard gelatin capsules for oral use. The dose was 750 mg once daily.
  Arms: Ceritinib
Drug: Pemetrexed — Pemetrexed was one of the chemotherapy treatments. Pemetrexed, a reconstituted solution, was intravenously administered over 10 minutes at 500 mg/m^2 every 21 days.
  Arms: Chemotherapy
Drug: Docetaxel — Docetaxel was one of the chemotherapy treatments. Docetaxel, a reconstituted solution, was intravenously administered over 1 hour, at 75 mg/m^2 every 21 days.
  Arms: Chemotherapy

SUMMARY:
The primary purpose of the study was to compare the antitumor activity of LDK378 vs. chemotherapy in patients previously treated with chemotherapy (platinum doublet) and crizotinib. Patients in the chemotherapy arm were given the option to switch to LDK378 after confirmed progressive disease (PD), while also had the choice to continue with pemetrexed treatment.

DETAILED DESCRIPTION:
A total of 231 patients were randomized to one of the two treatment arms in a 1:1 ratio. Randomization was stratified by World Health Organization (WHO) performance status (0 versus 1-2) and whether the patient had brain metastases at screening. The study was planned to be ended once the final overall survival (OS) analysis was performed (at the earliest of approximately 196 deaths observed or statistical significance reached at earlier OS interim analysis).

Following an agreement between Novartis and European Medicines Agency (EMA) in May 2023 to terminate the trial earlier, this study was completed when the total number of deaths was 190. Patients who had Response Evaluation Criteria In Solid Tumors (RECIST)-defined disease progression as confirmed by the Blinded Independent Review Committee (BIRC), but who, in the opinion of the Investigator, had continued clinical benefit from study treatment on either the chemotherapy arm or the ceritinib arm, continued to receive treatment. These patients continued assessments in the treatment phase. In addition, only patients randomized to the chemotherapy arm were allowed to crossover to receive ceritinib therapy (extension treatment [ET] phase) after BIRC-confirmed, RECIST-defined disease progression, and provided they met the eligibility requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC) that is anaplastic lymphoma kinase (ALK) positive as assessed by the FDA approved Abbott FISH Test.
2. Patient has stage IIIB or IV diagnosis and must have received one or two prior regimens (including platinum- doublet) of cytotoxic chemotherapy for the treatment of locally advanced or metastatic NSCLC.
3. Patient has at least one measurable lesion as defined by RECIST 1.1. A previously irradiated site lesion may only be counted as a target lesion if there is clear sign of progression since the irradiation
4. Patients must have received previous treatment with crizotinib for the treatment of locally advanced or metastatic NSCLC.

Exclusion Criteria:

1. Patient with known hypersensitivity to any of the excipients of LDK378 (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate)
2. Patient with a history of severe hypersensitivity reaction to pemetrexed or docetaxel or any known excipients of these drugs.
3. Patient with symptomatic central nervous system (CNS) metastases who is neurologically unstable or has required increasing doses of steroids within the 2 weeks prior to screening to manage CNS symptoms.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (86):
- United States (13):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Memorial Cancer Institute, Hollywood, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - University Of Miami, Miami, Florida
  - Loyola University Medical Center, Marywood, Illinois
  - Uni Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Sugarland, Sugar Land, Texas
  - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (9):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Suresnes
- Germany (8):
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Pokfulam
- Ireland (2):
  - Novartis Investigative Site, Limerick, Co Limerick
  - Novartis Investigative Site, Dublin
- Israel (2):
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
- Italy (10):
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Verona, VR
- Japan (11):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Niigata
- Novartis Investigative Site, El Achrafiyé, Lebanon
- Novartis Investigative Site, Groningen, Netherlands
- Novartis Investigative Site, Lisbon, Portugal
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Moscow Region Istra Village
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Spain (6):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Sankt Gallen
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Pendik Istanbul, Turkey
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
- United Kingdom (5):
  - Novartis Investigative Site, Cheltenham, Gloucestershire
  - Novartis Investigative Site, Aberdeen, Grampian Region
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kiura K, Imamura F, Kagamu H, Matsumoto S, Hida T, Nakagawa K, Satouchi M, Okamoto I, Takenoyama M, Fujisaka Y, Kurata T, Ito M, Tokushige K, Hatano B, Nishio M. Phase 3 study of ceritinib vs chemotherapy in ALK-rearranged NSCLC patients previously treated with chemotherapy and crizotinib (ASCEND-5): Japanese subset. Jpn J Clin Oncol. 2018 Apr 1;48(4):367-375. doi: 10.1093/jjco/hyy016. PMID 29474558
- [Derived] Shaw AT, Kim TM, Crino L, Gridelli C, Kiura K, Liu G, Novello S, Bearz A, Gautschi O, Mok T, Nishio M, Scagliotti G, Spigel DR, Deudon S, Zheng C, Pantano S, Urban P, Massacesi C, Viraswami-Appanna K, Felip E. Ceritinib versus chemotherapy in patients with ALK-rearranged non-small-cell lung cancer previously given chemotherapy and crizotinib (ASCEND-5): a randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2017 Jul;18(7):874-886. doi: 10.1016/S1470-2045(17)30339-X. Epub 2017 Jun 9. PMID 28602779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the following countries (with number of sites): Belgium (4), Canada (1), France (9), Germany (8), Hong Kong (3), Ireland (2), Israel (2), Italy (10), Japan (12), Republic of Korea (5), Lebanon (1), Netherlands (2), Portugal (1), Russia (3), Singapore (2), Spain (11), Switzerland (2), Turkey (3), United Kingdom (5), United States (13).
Pre-assignment Details: In the treatment phase, patients were randomized 1:1 to one of the treatment arms (ceritinib or chemotherapy). In the extension treatment phase, only patients randomized to the chemotherapy arm were allowed to crossover to receive ceritinib therapy after BIRC-confirmed, RECIST-defined disease progression.
Groups:
- Chemotherapy/Ceritinib: Patients randomized to chemotherapy who crossed over to ceritinib at the extension treatment phase
Period: Treatment Phase
Arm/Group | Ceritinib | Chemotherapy | Chemotherapy/Ceritinib
Started (Full Analysis Set: all patients to whom study treatment was assigned by randomization) | 115 | 116 | 0
Safety Set (All patients who received at least one dose of study drug) | 115 | 113 | 0
Completed (Patients who did not discontinue treatment at the end of the treatment phase) | 0 | 0 | 0
Not Completed | 115 | 116 | 0
Not completed — Adverse Event | 7 | 8 | 0
Not completed — Death | 9 | 5 | 0
Not completed — No longer required treatment | 0 | 1 | 0
Not completed — Physician Decision | 6 | 7 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Progressive disease | 79 | 87 | 0
Not completed — Study terminated by sponsor | 1 | 0 | 0
Not completed — Subject/guardian decision | 12 | 8 | 0
Period: Extension Treatment Phase
Arm/Group | Ceritinib | Chemotherapy | Chemotherapy/Ceritinib
Started (Patients randomized to chemotherapy who crossed over to the ceritinib arm) | 0 | 0 | 79
Crossover Analysis Set (Patients who crossed over to the ceritinib arm and received at least one dose of ceritinib) | 0 | 0 | 78
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 79
Not completed — Adverse Event | 0 | 0 | 6
Not completed — Death | 0 | 0 | 17
Not completed — Physician Decision | 0 | 0 | 5
Not completed — Progressive disease | 0 | 0 | 46
Not completed — Study terminated by sponsor | 0 | 0 | 1
Not completed — Subject/guardian decision | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceritinib | Chemotherapy | Total
Number analyzed (Participants) | 115 | 116 | 231
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (11.96) | 54.4 (11.61) | 53.7 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 61 | 129
  Male | 47 | 55 | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 30 | 38 | 68
  Black | 0 | 1 | 1
  Caucasian | 81 | 68 | 149
  Other | 2 | 4 | 6
  Unknown | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Blinded Independent Review Committee (BIRC)
Description: PFS was defined as the time from the date of randomization to the date of the first radiologically documented disease progression or death due to any cause.
Time Frame: From the date of randomization to the date of first radiologically documented disease progression or death due to any cause up to approximately 24 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 115 | 116
months | 5.4 [4.1 to 6.9] | 1.6 [1.4 to 2.8]
Statistical Analysis 1: Comparison: Ceritinib vs Chemotherapy; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.36 to 0.67]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from date of randomization to date of death due to any cause.
Time Frame: Up to approximately 114 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 115 | 116
months | 17.7 [14.2 to 23.7] | 20.1 [11.9 to 31.2]

3. Secondary Outcome: Progression Free Survival (PFS) Per Investigator Assessment
Description: as for outcome 1
Time Frame: Up to approximately 84 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 115 | 116
months | 6.2 [4.4 to 7.9] | 1.6 [1.4 to 2.6]

4. Secondary Outcome: Overall Response Rate (ORR) Per BIRC
Description: ORR was defined as the percentage of participants with a best overall response defined as complete response (CR) or partial response (PR): (CR+PR) per Response Evaluation Criteria in Solid Tumors (RECIST), v. 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 54 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 115 | 116
percentage of participants | 40.9 [31.8 to 50.4] | 6.9 [3.0 to 13.1]

5. Secondary Outcome: Overall Response Rate (ORR) Per Investigator Assessment
Description: ORR was defined as the percentage of participants with a best overall response defined as complete response (CR) or partial response (PR): (CR+PR) per Response Evaluation Criteria in Solid Tumors (RECIST), v. 1.1. CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 93 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 115 | 116
percentage of participants | 44.3 [35.1 to 53.9] | 6.9 [3.0 to 13.1]

6. Secondary Outcome: Duration of Response (DOR) Per BIRC
Description: DOR defined as the time from the first documented response (CR or PR) to the first documented progression or death due to underlying cancer. CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 54 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Patients with confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 47 | 8
months | 7.6 [5.4 to 8.3] | 10.4 [3.5 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

7. Secondary Outcome: Duration of Response (DOR) Per Investigator Assessment
Description: as for outcome 6
Time Frame: Up to approximately 93 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Data are reported for responders only. Patients with confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 51 | 8
months | 6.7 [5.5 to 8.3] | 8.3 [2.8 to 69.9]

8. Secondary Outcome: Disease Control Rate (DCR) Per BIRC
Description: DCR was defined as the percentage of participants with best overall response of CR, PR, or stable disease (SD). CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 54 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 115 | 116
percentage of participants | 76.5 [67.7 to 83.9] | 37.9 [29.1 to 47.4]

9. Secondary Outcome: Disease Control Rate (DCR) Per Investigator Assessment
Description: as for outcome 8
Time Frame: Up to approximately 93 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 115 | 116
percentage of participants | 80.0 [71.5 to 86.9] | 39.7 [30.7 to 49.2]

10. Secondary Outcome: Time to Response (TTR) Per BIRC
Description: TTR was defined as the time from date of randomization to date of first documented response (CR or PR). CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 52 weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: weeks
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 47 | 8
weeks | 6.71 [4.9 to 52.3] | 9.64 [5.4 to 43.3]

11. Secondary Outcome: Time to Response (TTR) Per Investigator Assessment
Description: as for outcome 10
Time Frame: Up to approximately 45 weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: weeks
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 47 | 8
weeks | 6.43 [4.9 to 45.4] | 14.71 [6.3 to 36.4]

12. Secondary Outcome: Overall Intracranial Response Rate (OIRR) Per BIRC
Description: OIRR was defined as the ORR based on lesions in brain (target, nontarget lesions (and new lesions, if applicable) and calculated as the percentage of patients with a best overall confirmed response of CR or PR in the brain per modified RECIST 1.1 as assessed by BIRC neuroradiologist. CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 18 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Patients with measurable and/or nonmeasurable disease in the brain at baseline as per BIRC neuroradiology review.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 66 | 67
percentage of participants | 10.6 [4.4 to 20.6] | 3.0 [0.4 to 10.4]

13. Secondary Outcome: Intracranial Disease Control Rate (IDCR) Per BIRC
Description: IDCR was defined as the DCR based on lesions in brain (target, non-target lesions (and new lesions, if applicable) and calculated as the proportion of patients with a best overall response of CR or PR or SD (or non-CR/nonPD) in the brain per modified RECIST 1.1 as assessed by BIRC neuro-radiologist. CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 18 months
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 66 | 67
percentage of participants | 71.2 [58.7 to 81.7] | 53.7 [41.1 to 66.0]

14. Secondary Outcome: Duration of Intracranial Response (DOIR) Per BIRC
Description: DOIR was defined as the DOR based on lesions in brain (target, non-target lesions (and new lesions, if applicable) and calculated from the time of first documented response of CR or PR to the date of the first documented disease progression in the brain or death due to any cause per modified RECIST 1.1 as assessed by BIRC neuro-radiologist. CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 18 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization. Patients with measurable and/or nonmeasurable disease in the brain at baseline as per BIRC neuroradiology review. patients with measurable and/or non-measurable disease in the brain at baseline as per BIRC neuro-radiology review, and with confirmed intracranial CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 6 | 1
months | 8.3 [2.7 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 16.7 [NA to NA] — The lower and upper limits of 95% CI were not estimable due to the single data point.

15. Secondary Outcome: Least Squares Mean Scores on the European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC-QLQC30)
Description: The EORTC QLQ-C30 questionnaire contained 30 items and was composed of both multi-item scales and single item measures. These included five functional scales (physical, role, emotional, cognitive, and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact), and a global health status/quality of life (QoL) scale.
  All of the scales and single items ranged from 0 to 100. A high scale score represented a higher response level. Thus, a high score for a functional scale indicated a high/healthy level of functioning, a high score for the QoL indicated high QoL, but a high score for a symptom scale/single item indicated a high level of symptomatology/problems. Data from all collected time points were combined and presented using a repeated measures model for longitudinal data.
Time Frame: Screening and treatment phase up to 92 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 107 | 86
score on a scale
  Global Health Status/QoL n=106,85: number analyzed (Participants) | 106 | 85
  Global Health Status/QoL n=106,85 | 62.9 (1.13) | 63.2 (1.74)
  Physical Functioning n=107,86 | 80.5 (1.04) | 75.4 (1.52)
  Emotional Functioning n=106,86: number analyzed (Participants) | 106 | 86
  Emotional Functioning n=106,86 | 82.4 (1.01) | 80.7 (1.54)
  Social Functioning n=106,86: number analyzed (Participants) | 106 | 86
  Social Functioning n=106,86 | 76.7 (1.56) | 71.6 (2.31)
  Cognitive Functioning n=106,86: number analyzed (Participants) | 106 | 86
  Cognitive Functioning n=106,86 | 86.7 (0.91) | 84.5 (1.40)
  Role Functioning n=107,86 | 72.6 (1.30) | 68.7 (1.98)
  Fatigue n=107,86 | 31.1 (1.10) | 36.1 (1.69)
  Nausea and Vomiting n=107,86 | 17.2 (1.08) | 9.4 (1.69)
  Pain n=107,86 | 21.4 (1.22) | 24.2 (1.85)
  Dyspnea n=107,86 | 17.4 (1.03) | 24.0 (1.62)
  Insomnia n=107,86 | 18.9 (1.33) | 25.6 (2.05)
  Appetite Loss n=107,86 | 21.2 (1.33) | 13.9 (2.07)
  Constipation n=107,86 | 15.0 (1.31) | 15.0 (2.00)
  Diarrhea n=106,86: number analyzed (Participants) | 106 | 86
  Diarrhea n=106,86 | 29.3 (1.29) | 11.4 (2.02)
  Financial Difficulties n=104,85: number analyzed (Participants) | 104 | 85
  Financial Difficulties n=104,85 | 15.5 (1.41) | 19.7 (2.10)

16. Secondary Outcome: EORTC QLQ-LC13 Time to Definitive Deterioration
Description: The Lung Cancer module of the EORTC's quality of life questionnaire (EORTC QLQ-LC13) was used in conjunction with the EORTC QLQ-C30 and provided information on an additional 13 items specifically related to lung cancer. The lung cancer module incorporated one multi-item scale to assess dyspnea, and 9 single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All of the domain scores ranged from 0 to 100. A high score indicated a high level of symptoms. QLQ-LC13 time to definitive deterioration was defined as the time from randomization to the earliest date a patient shows a 10 point or higher increase from baseline in any of the ALCLC13 scores related to pain in chest, cough, or dyspnea (with no later change below this threshold), or death due to any cause. Each cycle was 21 days.
Time Frame: Screening and treatment phase up to 92 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 115 | 116
months | 13.4 [8.4 to 16.7] | 2.8 [1.0 to 5.6]

17. Secondary Outcome: Least Squares Mean Scores on the Lung Cancer Symptom Scale (LCSS)
Description: The LCSS patient scale uses a 24-hour recall period and contains nine items: six measuring major symptoms for lung cancer (appetite loss, fatigue, cough, dyspnea, hemoptysis, pain), and three summary items related to total symptom distress, normal activity status, and overall quality of life. The total scale used is a 100 mm visual analog scale to measure the intensity of patient responses, with zero corresponding to the lowest rating (best status) and 100 representing the highest rating (worst status). The total score was calculated as the mean of the 9 items. Data from all collected time points were combined and presented using a repeated measures model for longitudinal data.
Time Frame: Screening and treatment phase up to 92 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 107 | 85
millimeters
  LCSS Total Score n=106,82: number analyzed (Participants) | 106 | 82
  LCSS Total Score n=106,82 | 22.0 (0.87) | 26.3 (1.33)
  Appetite Loss n=107,85 | 28.0 (1.26) | 26.6 (1.99)
  Fatigue n=107,84: number analyzed (Participants) | 107 | 84
  Fatigue n=107,84 | 34.6 (1.33) | 39.2 (2.06)
  Cough n=107,84: number analyzed (Participants) | 107 | 84
  Cough n=107,84 | 11.5 (1.01) | 18.4 (1.56)
  Shortness of Breath n=107,85 | 18.2 (0.99) | 24.8 (1.56)
  Hemoptysis n=107,85 | 1.8 (0.34) | 2.2 (0.55)
  Pain n=107,85 | 18.2 (1.25) | 24.3 (1.92)
  Total Symptom Distress n=107,85 | 20.7 (1.26) | 24.6 (1.92)
  Normal Activity Status n=107,85 | 31.3 (1.47) | 36.8 (2.21)
  Overall Quality of Life n=106,84: number analyzed (Participants) | 106 | 84
  Overall Quality of Life n=106,84 | 33.1 (1.27) | 36.4 (1.94)
  LCSS Average Symptom Burden Index n=107,83: number analyzed (Participants) | 107 | 83
  LCSS Average Symptom Burden Index n=107,83 | 18.8 (0.77) | 22.9 (1.20)

18. Secondary Outcome: Least Squares Mean Scores on the EQ-5D-5L Index
Description: The EQ-5D descriptive classification consists of five dimensions of health: mobility, self-care, usual activities, anxiety/depression and pain/discomfort. Patients are requested to select the statement which best describes their condition on that day for each dimension. EQ-5D-5L index scores can range from -0.59 to 1, where 1 is the best possible health state. Data from all collected time points were combined and presented using a repeated measures model for longitudinal data.
Time Frame: Screening and treatment phase up to 92 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 107 | 88
score on a scale | 0.7837 (0.01039) | 0.7108 (0.01533)

19. Secondary Outcome: Least Squares Mean Scores on the EQ-5D Visual Analogue Scale (VAS)
Description: The EQ-5D descriptive classification consists of five dimensions of health: mobility, self-care, usual activities, anxiety/depression and pain/discomfort. Patients are requested to select the statement which best describes their condition on that day for each dimension. EQ VAS scores can range from 0 to 100, where 100 is the best possible health state. Data from all collected time points were combined and presented using a repeated measures model for longitudinal data.
Time Frame: Screening and treatment phase up to 92 months
Population: The Full Analysis Set (FAS) consisted of all patients to whom study treatment had been assigned by randomization.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 106 | 86
score on a scale | 71.8 (0.98) | 69.0 (1.45)

20. Secondary Outcome: Cmax for Ceritinib
Description: The observed maximum plasma concentration following administration
Time Frame: Cycle 1, Day 1 and Cycle 2, Day 1: pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose. Each cycle was 21 days.
Population: Participants in the pharmacokinetic (PK) analysis set who had extensive PK collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 4 | 0
ng/mL
  Cycle 1, Day 1 n=4,0 | 90.4 (49.8) |
  Cycle 2, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Cycle 2, Day 1 n=2,0 | 1170 (17.7) |

21. Secondary Outcome: Tmax for Ceritinib
Description: The time to reach peak or maximum concentration
Time Frame: Cycle 1, Day 1 and Cycle 2, Day 1: pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose. Each cycle was 21 days.
Population: Participants in the pharmacokinetic (PK) analysis set who had extensive PK collection.
Measure: Median (Full Range); unit: hours
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 4 | 0
hours
  Cycle 1, Day 1 n=4,0 | 6.03 [4.17 to 23.6] |
  Cycle 2, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Cycle 2, Day 1 n=2,0 | 7.15 [6.17 to 8.13] |

22. Secondary Outcome: Tlast for Ceritinib
Description: The time to last quantifiable concentration
Time Frame: Cycle 1, Day 1 and Cycle 2, Day 1: pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose. Each cycle was 21 days.
Population: Participants in the pharmacokinetic (PK) analysis set who had extensive PK collection.
Measure: Median (Full Range); unit: hours
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 4 | 0
hours
  Cycle 1, Day 1 n=4,0 | 24 [23.6 to 24.1] |
  Cycle 2, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Cycle 2, Day 1 n=2,0 | 23.9 [23.7 to 24.2] |

23. Secondary Outcome: AUC0-24h for Ceritinib
Description: The area under the plasma concentration-time curve calculated from time zero to 24 hours
Time Frame: Cycle 1, Day 1 and Cycle 2, Day 1: pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose. Each cycle was 21 days.
Population: Participants in the pharmacokinetic (PK) analysis set who had extensive PK collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 4 | 0
h*ng/mL
  Cycle 1, Day 1 n=4,0 | 1470 (65.1) |
  Cycle 2, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Cycle 2, Day 1 n=2,0 | 25000 (19.0) |

24. Secondary Outcome: Mean Accumulation Ratio (Racc) for Ceritinib
Description: Accumulation ratio calculated using AUC0-24 values obtained from a dosing interval at steady-state (Cycle 2, Day 1) divided by AUC0-24 on Cycle 1, Day 1.
Time Frame: Cycle 1, Day 1 and Cycle 2, Day 1: pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose. Each cycle was 21 days.
Population: Participants in the pharmacokinetic (PK) analysis set who had extensive PK collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 1 | 0
ratio
  Cycle 1, Day 1 n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 2, Day 1 n=1,0 | 15.5 (NA) — The geometric coefficient of variation was not estimable due to the single data point. |

25. Secondary Outcome: Clearance Rate at Steady State (CLss/F) for Ceritinib
Description: The apparent total body clearance from plasma. CLss/F is calculated from AUC0-24 assuming steady state (CLss/F=Dose/AUC0-24).
Time Frame: Cycle 1, Day 1 and Cycle 2, Day 1: pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose. Each cycle was 21 days.
Population: Participants in the pharmacokinetic (PK) analysis set who had extensive PK collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Ceritinib | Chemotherapy
Number analyzed (Participants) | 2 | 0
L/h
  Cycle 1, Day 1 n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 2, Day 1 n=2,0 | 30 (19.0) |

26. Secondary Outcome: Post-Hoc: All Collected Deaths
Description: Pre-treatment deaths: from day of patient's informed consent to the day before first dose of study treatment. On-treatment deaths: from first dose of study treatment to 30 days following the last dose of study treatment at the end of treatment phase. For crossover patients, from first dose of ceritinib at the extension treatment phase to 30 days following the last dose. Survival Follow-up deaths: from Day 31 after last dose of study treatment to the data cut-off date.
Time Frame: Pre-treatment and on-treatment deaths: Up to approximately 8 years. Post-treatment survival follow-up deaths: Up to an additional 2.5 years.
Population: The analysis included patients who received at least one dose of study drug. For the Chemotherapy/Ceritinib group, the analysis included patients randomized to the chemotherapy arm who crossed over to receive at least one dose of ceritinib in the extension-treatment phase. For pre-treatment deaths, all randomized patients are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceritinib | Chemotherapy | Chemotherapy/Ceritinib
Number analyzed (Participants) | 115 | 116 | 78
Participants
  Pre-treatment deaths: number analyzed (Participants) | 115 | 116 | 0
  Pre-treatment deaths | 0 | 2 | 0
  On-treatment deaths: number analyzed (Participants) | 115 | 113 | 78
  On-treatment deaths | 16 | 5 | 19
  Survival follow-up deaths: number analyzed (Participants) | 93 | 23 | 55
  Survival follow-up deaths | 86 | 18 | 44
  All deaths | 102 | 25 | 63

ADVERSE EVENTS:
Time Frame: From day of first dose of study medication to last dose of study medication plus 30 days, up to approximately 8 years. Deaths were also collected in the survival follow-up phase from 31 days after last dose of study medication until the end of the study, up to approximately 2.5 additional years. These were not considered AEs.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival included participants who entered the survival follow-up period. In the on-treatment and survival follow-up periods, patients were analyzed according to the treatment received. Serious and non-serious adverse events were not assessed in the pre-treatment arms/groups.
Groups:
- Ceritinib (Pre-treatment); Ceritinib (On-treatment); Ceritinib (Survival Follow-up): Ceritinib 750 mg
- Chemotherapy (Pre-treatment); Chemotherapy (On-treatment); Chemotherapy (Survival Follow-up): Chemotherapy as determined by BIRC
- Chemotherapy/Ceritinib (Pre-treatment); Chemotherapy/Ceritinib (On-treatment); Chemotherapy/Ceritinib (Survival Follow-up): Patients randomized to chemotherapy who crossed over to ceritinib at the extension treatment phase
Arm/Group | Ceritinib (Pre-treatment) | Chemotherapy (Pre-treatment) | Chemotherapy/Ceritinib (Pre-treatment) | Ceritinib (On-treatment) | Chemotherapy (On-treatment) | Chemotherapy/Ceritinib (On-treatment) | Ceritinib (Survival Follow-up) | Chemotherapy (Survival Follow-up) | Chemotherapy/Ceritinib (Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 0/115 | 2/116 | 0/0 | 16/115 | 5/113 | 19/78 | 86/93 | 18/23 | 44/55
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 57/115 | 35/113 | 45/78 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 114/115 | 111/113 | 76/78 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceritinib (Pre-treatment) (N=0) | Chemotherapy (Pre-treatment) (N=0) | Chemotherapy/Ceritinib (Pre-treatment) (N=0) | Ceritinib (On-treatment) (N=115) | Chemotherapy (On-treatment) (N=113) | Chemotherapy/Ceritinib (On-treatment) (N=78) | Ceritinib (Survival Follow-up) (N=0) | Chemotherapy (Survival Follow-up) (N=0) | Chemotherapy/Ceritinib (Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Acute coronary syndrome (Cardiac disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | NA | NA | NA | 2 | 1 | 0 | NA | NA | NA
Atrial flutter (Cardiac disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Cardiac arrest (Cardiac disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Myocardial ischaemia (Cardiac disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Pericardial effusion (Cardiac disorders) | NA | NA | NA | 4 | 1 | 1 | NA | NA | NA
Pericarditis (Cardiac disorders) | NA | NA | NA | 1 | 0 | 1 | NA | NA | NA
Ventricular extrasystoles (Cardiac disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Lenticular opacities (Eye disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Visual field defect (Eye disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Colitis (Gastrointestinal disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | NA | NA | NA | 2 | 0 | 1 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | 1 | NA | NA | NA
Faecaloma (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Gastric perforation (Gastrointestinal disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Gastritis (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Gastrointestinal obstruction (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Gastrointestinal perforation (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Gastrointestinal toxicity (Gastrointestinal disorders) | NA | NA | NA | 1 | 0 | 1 | NA | NA | NA
Haematemesis (Gastrointestinal disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Large intestine perforation (Gastrointestinal disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Nausea (Gastrointestinal disorders) | NA | NA | NA | 8 | 0 | 4 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | NA | NA | NA | 6 | 0 | 5 | NA | NA | NA
Asthenia (General disorders) | NA | NA | NA | 2 | 3 | 2 | NA | NA | NA
Chest pain (General disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Condition aggravated (General disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Fatigue (General disorders) | NA | NA | NA | 2 | 1 | 1 | NA | NA | NA
General physical health deterioration (General disorders) | NA | NA | NA | 7 | 2 | 1 | NA | NA | NA
Multiple organ dysfunction syndrome (General disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Non-cardiac chest pain (General disorders) | NA | NA | NA | 2 | 0 | 3 | NA | NA | NA
Pain (General disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Pyrexia (General disorders) | NA | NA | NA | 4 | 2 | 1 | NA | NA | NA
Sudden death (General disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Acute hepatic failure (Hepatobiliary disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Hepatic lesion (Hepatobiliary disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Jaundice (Hepatobiliary disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Bacteraemia (Infections and infestations) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Bacterial pyelonephritis (Infections and infestations) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Biliary tract infection (Infections and infestations) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Bronchitis (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Hepatic infection (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Infection (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Localised infection (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | NA | NA | NA | 1 | 0 | 1 | NA | NA | NA
Mucosal infection (Infections and infestations) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Neutropenic sepsis (Infections and infestations) | NA | NA | NA | 0 | 2 | 0 | NA | NA | NA
Oral herpes (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Oropharyngeal candidiasis (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Pneumonia (Infections and infestations) | NA | NA | NA | 6 | 4 | 6 | NA | NA | NA
Pseudomembranous colitis (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Respiratory tract infection (Infections and infestations) | NA | NA | NA | 3 | 0 | 1 | NA | NA | NA
Typhoid fever (Infections and infestations) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Urosepsis (Infections and infestations) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Viral infection (Infections and infestations) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Radius fracture (Injury, poisoning and procedural complications) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Tracheal obstruction (Injury, poisoning and procedural complications) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
C-reactive protein increased (Investigations) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Electrocardiogram T wave inversion (Investigations) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Neutrophil count decreased (Investigations) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | NA | NA | NA | 1 | 1 | 0 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | NA | NA | NA | 2 | 1 | 0 | NA | NA | NA
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | NA | NA | NA | 1 | 0 | 3 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | NA | NA | NA | 1 | 0 | 1 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | NA | NA | NA | 1 | 0 | 1 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 1 | 2 | 1 | NA | NA | NA
Mobility decreased (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 2 | 0 | 1 | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | NA | 1 | 1 | 0 | NA | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | NA | 0 | 0 | 2 | NA | NA | NA
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Aphasia (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Brain oedema (Nervous system disorders) | NA | NA | NA | 1 | 1 | 1 | NA | NA | NA
Cerebellar infarction (Nervous system disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Cognitive disorder (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Coordination abnormal (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Depressed level of consciousness (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Epilepsy (Nervous system disorders) | NA | NA | NA | 2 | 0 | 0 | NA | NA | NA
Headache (Nervous system disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Intracranial mass (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Loss of consciousness (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Paraesthesia (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Paraparesis (Nervous system disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Parkinsonism (Nervous system disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Partial seizures (Nervous system disorders) | NA | NA | NA | 1 | 0 | 1 | NA | NA | NA
Petit mal epilepsy (Nervous system disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Presyncope (Nervous system disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Seizure (Nervous system disorders) | NA | NA | NA | 1 | 2 | 2 | NA | NA | NA
Syncope (Nervous system disorders) | NA | NA | NA | 1 | 1 | 0 | NA | NA | NA
Device failure (Product Issues) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Anxiety (Psychiatric disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Anxiety disorder (Psychiatric disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Confusional state (Psychiatric disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Hallucination (Psychiatric disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Mental status changes (Psychiatric disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Renal failure (Renal and urinary disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Urinary bladder rupture (Renal and urinary disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Urinary retention (Renal and urinary disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 8 | 5 | 4 | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 1 | 0 | NA | NA | NA
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 5 | 2 | 5 | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 | 1 | 0 | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 | 0 | 2 | NA | NA | NA
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 1 | 0 | 0 | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 3 | 0 | 2 | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | NA | NA | NA | 1 | 0 | 1 | NA | NA | NA
Lymphoedema (Vascular disorders) | NA | NA | NA | 0 | 0 | 1 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceritinib (Pre-treatment) (N=0) | Chemotherapy (Pre-treatment) (N=0) | Chemotherapy/Ceritinib (Pre-treatment) (N=0) | Ceritinib (On-treatment) (N=115) | Chemotherapy (On-treatment) (N=113) | Chemotherapy/Ceritinib (On-treatment) (N=78) | Ceritinib (Survival Follow-up) (N=0) | Chemotherapy (Survival Follow-up) (N=0) | Chemotherapy/Ceritinib (Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | NA | NA | NA | 7 | 20 | 8 | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | NA | NA | NA | 0 | 6 | 0 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | NA | NA | NA | 3 | 9 | 6 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | NA | NA | NA | 6 | 25 | 6 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | NA | NA | NA | 29 | 10 | 20 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | NA | NA | NA | 22 | 5 | 11 | NA | NA | NA
Constipation (Gastrointestinal disorders) | NA | NA | NA | 25 | 15 | 20 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | NA | NA | NA | 84 | 21 | 57 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | NA | NA | NA | 6 | 1 | 2 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | NA | NA | NA | 3 | 3 | 4 | NA | NA | NA
Nausea (Gastrointestinal disorders) | NA | NA | NA | 73 | 27 | 46 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | NA | NA | NA | 8 | 15 | 5 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | NA | NA | NA | 61 | 9 | 37 | NA | NA | NA
Asthenia (General disorders) | NA | NA | NA | 29 | 19 | 13 | NA | NA | NA
Fatigue (General disorders) | NA | NA | NA | 34 | 32 | 17 | NA | NA | NA
Malaise (General disorders) | NA | NA | NA | 7 | 5 | 7 | NA | NA | NA
Non-cardiac chest pain (General disorders) | NA | NA | NA | 16 | 4 | 11 | NA | NA | NA
Oedema peripheral (General disorders) | NA | NA | NA | 6 | 11 | 5 | NA | NA | NA
Pain (General disorders) | NA | NA | NA | 8 | 2 | 5 | NA | NA | NA
Pyrexia (General disorders) | NA | NA | NA | 19 | 16 | 14 | NA | NA | NA
Bronchitis (Infections and infestations) | NA | NA | NA | 4 | 4 | 4 | NA | NA | NA
Cystitis (Infections and infestations) | NA | NA | NA | 0 | 0 | 4 | NA | NA | NA
Influenza (Infections and infestations) | NA | NA | NA | 7 | 1 | 2 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | NA | NA | NA | 13 | 2 | 6 | NA | NA | NA
Oral candidiasis (Infections and infestations) | NA | NA | NA | 6 | 3 | 1 | NA | NA | NA
Pneumonia (Infections and infestations) | NA | NA | NA | 6 | 1 | 5 | NA | NA | NA
Respiratory tract infection (Infections and infestations) | NA | NA | NA | 7 | 1 | 3 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | NA | NA | NA | 3 | 4 | 5 | NA | NA | NA
Urinary tract infection (Infections and infestations) | NA | NA | NA | 1 | 4 | 6 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | NA | NA | NA | 52 | 10 | 29 | NA | NA | NA
Amylase increased (Investigations) | NA | NA | NA | 7 | 3 | 5 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | NA | NA | NA | 44 | 5 | 25 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | NA | NA | NA | 28 | 1 | 12 | NA | NA | NA
Blood creatinine increased (Investigations) | NA | NA | NA | 24 | 1 | 21 | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | NA | NA | NA | 14 | 0 | 8 | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | NA | NA | NA | 27 | 3 | 18 | NA | NA | NA
Lipase increased (Investigations) | NA | NA | NA | 1 | 0 | 5 | NA | NA | NA
Neutrophil count decreased (Investigations) | NA | NA | NA | 1 | 8 | 0 | NA | NA | NA
Weight decreased (Investigations) | NA | NA | NA | 37 | 7 | 13 | NA | NA | NA
White blood cell count decreased (Investigations) | NA | NA | NA | 2 | 7 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | NA | NA | NA | 50 | 23 | 25 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | NA | NA | NA | 9 | 3 | 5 | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | NA | NA | NA | 4 | 2 | 5 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | NA | NA | NA | 12 | 1 | 7 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 23 | 16 | 13 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 27 | 9 | 10 | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 4 | 5 | 5 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 11 | 4 | 3 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 6 | 14 | 6 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 8 | 2 | 1 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 8 | 7 | 4 | NA | NA | NA
Dizziness (Nervous system disorders) | NA | NA | NA | 13 | 8 | 10 | NA | NA | NA
Headache (Nervous system disorders) | NA | NA | NA | 28 | 18 | 16 | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | NA | NA | NA | 2 | 9 | 1 | NA | NA | NA
Paraesthesia (Nervous system disorders) | NA | NA | NA | 3 | 6 | 0 | NA | NA | NA
Somnolence (Nervous system disorders) | NA | NA | NA | 5 | 3 | 5 | NA | NA | NA
Tremor (Nervous system disorders) | NA | NA | NA | 6 | 0 | 7 | NA | NA | NA
Anxiety (Psychiatric disorders) | NA | NA | NA | 4 | 5 | 7 | NA | NA | NA
Insomnia (Psychiatric disorders) | NA | NA | NA | 11 | 13 | 6 | NA | NA | NA
Pollakiuria (Renal and urinary disorders) | NA | NA | NA | 0 | 2 | 4 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 20 | 20 | 13 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 18 | 18 | 13 | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 | 6 | 0 | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 5 | 4 | 4 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 2 | 4 | 7 | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 7 | 7 | 6 | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 2 | 6 | 2 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | NA | NA | NA | 6 | 24 | 2 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | NA | NA | NA | 6 | 2 | 4 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | NA | NA | NA | 14 | 7 | 6 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | NA | NA | NA | 15 | 13 | 15 | NA | NA | NA
Hypertension (Vascular disorders) | NA | NA | NA | 4 | 4 | 5 | NA | NA | NA

LIMITATIONS AND CAVEATS:
Although 116 patients were randomized to the Chemotherapy arm, 3 did not receive study drug and were excluded from the Safety set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.